CLINICAL TRIAL: NCT00314873
Title: Pilot Study of Imatinib (Gleevec) as Treatment for Advanced Thymic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603-21/ IUCRO-0147
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Thymic Carcinoma
Keywords: Thymic malignancy; Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Gleevec (imatinib) — Imatinib 600mg po qd X 21 days.

SUMMARY:
This study is important to demonstrate if single agent activity is noted for patients with thymic tumors over expressing c-kit and/or PDGF. If this current trial is positive, it opens the door to evaluate other combination of drugs with imatinib in thymic tumors.

DETAILED DESCRIPTION:
Thymic carcinomas are particularly more concerning due to their aggressive metastatic nature and shorter overall survival, in comparison to their lesser-malignant thymoma counterparts. This necessitates the need for systemic therapy. Due to the paucity of thymic carcinoma cases, the ideal regimen for locally advanced or metastatic thymic carcinomas is not defined.To this point, there has not been a study using imatinib in thymic tumors expressing the KIT tyrosine kinase protein or PDGF tyrosine kinase protein. This study is important to demonstrate if single agent activity is noted for patients with thymic tumors over expressing c-kit and/or PDGF. If this current trial is positive, it opens the door to evaluate other combination of drugs with imatinib in thymic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of advanced C-KIT positive or PDGFR positive thymic carcinoma. For protocol purposes, advanced disease is defined as disease
* Patient must have at least one documented measurable lesion obtained by imaging within 28 days prior to being registered for protocol therapy.
* No prior imatinib therapy.
* Age > 18 years at the time of consent
* ECOG performance status of 0 or 1
* ANC ≥ 1500/mm3,Platelet count ≥ 100,000/mm,Total bilirubin < 1.5ULN,3.10 Serum creatinine ≤ 1.7 mg/dl,ALT and AST ≤ 3 x ULN

Exclusion Criteria:

* Clinically significant infections as judged by the treating investigator
* Clinically significant concurrent illnesses
* Females of childbearing potential not using birth control or breastfeeding
* Prior radiation therapy > 25% of the bone marrow
* Symptomatic brain metastasis
* History of Grade III/IV cardiac problems
* History of major surgery within 14 days prior to being registered
* Treatment with any investigational agent within 30 days prior to being registered for protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate of imatinib in patients with c-kit or PDGF positive thymic carcinoma. | baseline through progression
To determine the duration of remission of patients with thymic carcinoma treated with imatinib. | baseline through progression
To determine the toxicity of imatinib in this patient population. | baseline through end of study
To determine the incidence of kit mutations in thymic malignancies. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Loehrer, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States